CLINICAL TRIAL: NCT00993629
Title: Adjunctive Pregnenolone in PTSD and Depression in OEF/OIF Veterans
Brief Title: Adjunctive Pregnenolone in Post-Traumatic Stress Disorder (PTSD) and Depression in Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) Veterans
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI turned down funding.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B7064-W
Record Dates: First submitted 2009-10-07; First posted 2009-10-12 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Post-traumatic Stress Disorder; Major Depressive Disorder
Keywords: PTSD; Depression; Neurosteroids
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Depression | interventions — Pregnenolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): adjunctive pregnenolone
  Interventions: Drug: pregnenolone
- Arm 2 (Placebo Comparator): adjunctive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregnenolone — Administered adjunctively to "treatment as usual"
  Arms: Arm 1
Drug: placebo — adjunctive placebo
  Arms: Arm 2

SUMMARY:
This study will be an 8-week randomized, placebo-controlled clinical trial of pregnenolone administered adjunctively to treatment as usual in PTSD and depression in OEF/OIF Veterans.

DETAILED DESCRIPTION:
PTSD and depression are critical areas of immediate impact to Operation Enduring Freedom and Operation Iraqi Freedom (OEF/OIF) Veterans. Current treatments for PTSD (which frequently co-occurs with depression) remain limited, with many patients remaining symptomatic despite single or combination administration of SSRIs, mood stabilizers, antipsychotics and sedatives/hypnotics. In addition, many patients treated for depression remain symptomatic. New interventions are thus urgently needed in PTSD with co-occurring depression to ensure optimal functional outcomes for our Service members and their families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD,
* diagnosis of MDD,
* age 18-55,
* no change in psychotropic medication for >=4 weeks,
* no anticipated need to to alter psychotropic medication for duration of study

Exclusion Criteria:

* Unstable medical/neurological illness,
* diagnosis of bipolar disorder, schizophrenia or other psychotic disorder,
* cognitive disorder,
* substance dependence,
* positive urine drug screen at screening,
* use of hormonal supplementation,
* pregnancy/lactation,
* female patients who are sexually active and not using acceptable non-hormonal birth control,
* initiation/change of psychotherapy within 3 months of randomization,
* recent/current electroconvulsive therapy,
* regular use of opiates/barbiturates/benzodiazepines

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victoria M Payne, MD MS, Principal Investigator — VA Medical Center, Durham
Locations (1):
- VA Medical Center, Durham, Durham, North Carolina, United States